CLINICAL TRIAL: NCT03665220
Title: Effects of Two Home Ergonomics Programmes on Post-stroke Patients' Quality of Life and Functional Capacity: a Randomised Controlled Clinical Trial
Brief Title: Effects of Two Home Ergonomics Programmes in Post-stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, José Manuel Pérez Mármol, Principal Investigator, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Rehab in post-stroke patients
Record Dates: First submitted 2018-09-06; First posted 2018-09-11 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Stroke; Quality of Life
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ergonomic adjustment group (Experimental): Ergonomic intervention program at home for post-stroke patients. The ergonomic adjustments made were based on a prior assessment of the patient's needs in this respect, using a purpose-made home inspection form.
  Interventions: Other: Ergonomic adjustments
- Kinesiotherapy + ergonomics group (Experimental): A Kinesiotherapy plus ergonomic adjustments program for post-stroke patients. This group received, in addition to the ergonomic adjustments described above, sessions of postural orientation and kinesiotherapy (therapeutic exercises).
  Interventions: Other: Kinesiotherapy plus ergonomic adjustments
- Healthcare education (Active Comparator): A conservative intervention program for post-stroke patients
  Interventions: Other: Healthcare education

INTERVENTIONS:
Other: Ergonomic adjustments — The ergonomic adjustments made were based on a prior assessment of the patient's needs in this respect, using a purpose-made home inspection form .
  Arms: Ergonomic adjustment group
Other: Kinesiotherapy plus ergonomic adjustments — This group received, in addition to the ergonomic adjustments described above, sessions of postural orientation and kinesiotherapy (therapeutic exercises).
  Arms: Kinesiotherapy + ergonomics group
Other: Healthcare education — This group received health education information, based on an illustrated manual with advice for patients with chronic stroke.
  Arms: Healthcare education

SUMMARY:
The main objective of the clinical trial is to evaluate the effectiveness of two home ergonomics programmes, by reference to a control group, on functional capacity and quality of life in post-stroke patients.

DETAILED DESCRIPTION:
For post-stroke patients, rehabilitation must address different aspects. When the resulting condition has become established, treatment should take the form of a mixed intervention model, incorporating preventive, rehabilitational and compensatory or adaptive approaches, aimed at enhancing the patient's performance within the environment. Physiotherapy and occupational therapy are key disciplines in the composition of multi- and inter-disciplinary teams for the care of stroke patients. In this clinical trial we evaluate the effectiveness of two programmes of ergonomic intervention in the home, with respect to levels of functionality (performance of activities of daily living) and the quality of life of post-stroke patients, by reference to a control group.

ELIGIBILITY:
Inclusion Criteria:

* stroke diagnosed 6-24 months previously
* aged over 18 years
* ability to speak and understand Portuguese.

Exclusion Criteria:

* severe cognitive deficit
* severe aphasia
* other associated neurological disease
* musculoskeletal pathology
* drug or alcohol abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
Change from the World Health Organization's Quality of Life Questionnaire (WhoQol-Bref) at 12 weeks | Twelve weeks
  The quality of life is assessed on the WHOQoL-Bref scale, on a range from 0 to 100 points, where 100 is the highest level of quality of life. For each domain, with the exception of the first two questions, the quality of life was considered to be impaired when a score <70 points was assigned.
Change from the World Health Organization's Quality of Life Questionnaire (WhoQol-Bref) at 24 weeks | Twenty four weeks
  The quality of life is assessed on the WHOQoL-Bref scale, on a range from 0 to 100 points, where 100 is the highest level of quality of life. For each domain, with the exception of the first two questions, the quality of life was considered to be impaired when a score <70 points was assigned.

SECONDARY OUTCOMES:
Change from the Older Americans Resources and Services (OARS) scale at 12 weeks | Twelve weeks
  Functional capacity is measured using the Older Americans Resources and Services (OARS) scale, which consists of two parts. The Brazilian-language version of this scale allows each part to be used independently. Each item is scored according to a Likert scale, ranging from 0 to 2 points, where 0 indicates a total level of dependence for the performance of ADL, 1 point corresponds to partial independence, and 2 points represents a satisfactory level of independence. The scale consists of 15 items that evaluate activities such as using the telephone, transport, shopping, preparing and consuming food, cleaning and housework, administering medicines, financial affairs, dressing and undressing, personal hygiene and grooming, functional mobility, getting into and out of bed, bathing and mobility in the bathroom.
Change from the Older Americans Resources and Services (OARS) scale at 24 weeks | Twenty four weeks
  Functional capacity is measured using the Older Americans Resources and Services (OARS) scale, which consists of two parts. The Brazilian-language version of this scale allows each part to be used independently. Each item is scored according to a Likert scale, ranging from 0 to 2 points, where 0 indicates a total level of dependence for the performance of ADL, 1 point corresponds to partial independence, and 2 points represents a satisfactory level of independence. The scale consists of 15 items that evaluate activities such as using the telephone, transport, shopping, preparing and consuming food, cleaning and housework, administering medicines, financial affairs, dressing and undressing, personal hygiene and grooming, functional mobility, getting into and out of bed, bathing and mobility in the bathroom.

CONTACTS AND LOCATIONS:
Overall Officials: José Manuel Pérez Mármol, Principal Investigator — Department of Physiotherapy. Faculty of Health Sciences, University of Granada
Locations (1):
- José Manuel Pérez Mármol, Granada, Spain